CLINICAL TRIAL: NCT01133912
Title: Phase Ib Study of Preoperative Chemotherapy With Paclitaxel, Gemcitabine, and Lapatinib (Tykerb®) (PGT) in Patients With HER2 Positive Operable Breast Cancer
Brief Title: Preoperative Chemotherapy With Paclitaxel, Gemcitabine, and Lapatinib (Tykerb®) (PGT)
Acronym: PGT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jungsil Ro (Other Government)
Collaborators: GlaxoSmithKline (Industry); HK inno.N Corporation (Industry)
Responsible Party: Sponsor-Investigator, Jungsil Ro, Chief, Center for Clinical Trials, National Cancer Center, Korea, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-08-370
Record Dates: First submitted 2010-02-17; First posted 2010-05-31 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: Patients with HER2 Positive Operable Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Gemcitabine; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paclitaxel, gemcitabine, lapatinib (Experimental): paclitaxel 80mg/m2 D1, D8 gemcitabine 1000mg/m2 D1, D8, every 3 weeks, 6 cycle lapatinib(Tykerb®)1000mg every day
  Interventions: Drug: paclitaxel, gemcitabine, lapatinib

INTERVENTIONS:
Drug: paclitaxel, gemcitabine, lapatinib — Patients receive paclitaxel and gemcitabine intravenously (iv) on day 1 and 8, and oral lapatinib once daily. Lapatinib with fixed dose will be given once a day p.o. from day 1 without resting during each cycle. The starting doses of paclitaxel 80mg/m2 and gemcitabine 1000mg/m2 iv, on day 1 and 8, and lapatinib 1000mg p.o., daily (dose level 1) will be administered every 21 days.
  Other Names: Paclitaxel; Gemzar; Tykerb

SUMMARY:
Primary objectives :

1. To evaluate the recommended dose of the combination of paclitaxel, gemcitabine, and lapatinib (Tykerb®) (PGT) as preoperative chemotherapy in patients with HER2 positive operable breast cancer

Secondary objectives :

1. To evaluate the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of PGT
2. To determine the safety profile
3. To assess pCR in primary tumor and axillary LN
4. To evaluate clinical response rate, disease free survival (DFS), and overall survival (OS)
5. To assess breast conserving rate after preoperative PGT

DETAILED DESCRIPTION:
Unlike adjuvant chemotherapy, primary (preoperative) chemotherapy will shrink tumor and allow some patients to become candidates for conservative surgery and avoid mastectomy. It also is an in vivo chemosensitivity test and the result is a predictive marker for clinical outcomes. Paclitaxel is a highly active antitumor agent that promotes microtubule assembly by binding to tubulin and inhibiting depolymerization. Paclitaxel has been shown to be an effective agent in the treatment of breast cancer. Gemcitabine is a cytosine arabinoside prodrug analog and shows response rates of 15% to 46% as a single agent with very low toxicity. The combination of gemcitabine and paclitaxel is valuable because of the different mechanisms of action of each drug and their non-overlapping toxicities. Phase II studies of paclitaxel plus gemcitabine in anthracycline-pretreated metastatic breast cancer showed good tolerance and encouraging response rates (40%-55%). Paclitaxel plus gemcitabine combination showed overall survival benefit compared to paclitaxel alone in patients with metastatic breast cancer in an interim overall survival report. A phase II study with preoperative paclitaxel and gemcitabine in stage II/III showed 18 % pCR rate at NCC (ASCO 2007 abstract #11080) In HER2 positive breast cancer, HER2 targeted therapies with trastuzumab and lapatinib have shown much improved clinical response in palliative setting. It also showed that adding trastuzumab to sequential paclitaxel and FEC chemotherapy significantly increased pCR (25% vs 66.7%) in preoperative setting for HER2 positive disease. Recently, paclitaxel, gemcitabine, and trastuzumab combination (PGH) for 6 cycles in patients with HER2 positive and node positive operable breast cancer observed a strikingly high pCR rate in both tumor and LN in an interim analysis of multicenter phase II preoperative study in Korea (28 of 47 (61%)). Lapatinib (Tykerb®), a dual tyrosine kinase inhibitor of ErbB1 and HER2 signaling pathways and it has shown to inhibit the growth of HER2 overexpressing breast cancer cells that do not respond to trastuzumab after long-term conditioning. We will examine the hypothesis that paclitaxel, gemcitabine, and lapatinib (Tykerb®) (PGT) combination could improve the pathological complete response rate of HER2 positive breast cancer when applied as a preoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and newly diagnosed operable breast cancer
* Documented HER2 positive disease : 3+ overexpression by IHC or HER2 gene amplification by FISH
* ECOG performance status 0-2
* Age ≥ 18 years
* Clinical stage II or III operable breast cancer
* Axillary node positivity determined by cytology
* No prior hormonal, chemotherapy, or radiotherapy is allowed
* No breast operation other than biopsy to make diagnosis is allowed
* Negative urine pregnancy test within 7 days prior to registration in premenopausal patients
* Adequate hematopoietic function: Absolute granulocyte count ≥1,500/mm3, platelet ≥100,000/mm3, hemoglobin ≥10g/mm3
* Adequate hepatic function: total bilirubin ≤1.5mg/dL, AST/ALT ≤2 x UNL, alkaline phosphatase ≤2 x UNL
* Adequate renal function: Serum creatinine ≤1.5mg/dL
* Adequate cardiac function:

  1. Normal or nonspecific EKG taken within 1 month of enrollment
  2. LVEF ≥50% by MUGA or echocardiogram taken within 4 weeks of enrollment
* Ability to understand and comply with protocol during study period
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Pregnant or lactating women
* Patients who received hormonal, chemotherapy or radiotherapy for breast cancer
* Patients with bilateral breast cancer
* Patients who underwent surgery for breast cancer
* Patients with node-negative stage IIA (T2N0) breast cancer
* Patients who have history of cancer other than in situ uterine cervix cancer or nonmelanotic skin cancer
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled GI disease (e.g., Crohn's disease, ulcerative colitis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the recommended dose of the combination of paclitaxel, gemcitabine, and lapatinib (Tykerb®) (PGT) as preoperative chemotherapy in patients with HER2 positive operable breast cancer | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, MD, Principal Investigator — National Cencer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea